CLINICAL TRIAL: NCT05120440
Title: The Effect of Breakfast Consumption on Afternoon Resistance Training Performance in Habitual Breakfast Consumers and Non-Consumers
Brief Title: The Effect of Breakfast Consumption on Afternoon Resistance Training Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB2021-649
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Resistance Training; Breakfast
Keywords: resistance training; breakfast; intermittent fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast Omission (Experimental): This arm will consist of omission of breakfast and consumption of standardized food items solely at lunch preceding afternoon resistance exercise.
  Interventions: Other: Breakfast omission
- Breakfast Consumption (Active Comparator): This arm will consist of consumption of standardized food items at breakfast and lunch preceding afternoon resistance exercise.
  Interventions: Other: Breakfast consumption

INTERVENTIONS:
Other: Breakfast omission — Breakfast omission will consist of not eating breakfast on the morning of afternoon resistance training performance assessment.
  Arms: Breakfast Omission
Other: Breakfast consumption — Breakfast consumption will consist of eating a standardized breakfast on the morning of afternoon resistance training performance assessment.
  Arms: Breakfast Consumption

SUMMARY:
This study is a randomized crossover trail examining the effect of breakfast consumption or omission on afternoon resistance training performance. Resistance-trained adults will complete a resistance training workout comprised of barbell back squat, barbell bench press, and barbell conventional deadlift following either consuming breakfast and lunch, or the same amount of food consumed solely at lunch. For each testing session the participants will be provided with all food to consume prior to arriving at the laboratory. Major performance outcomes will be total repetition volume completed for each exercise (i.e. bench press, squat, and deadlift) and the entire workout (each individual trial), along with barbell kinematics for each exercise.

DETAILED DESCRIPTION:
OVERVIEW

This study is a randomized crossover trail examining the effect of breakfast consumption or omission on afternoon resistance training performance. Resistance-trained adults will complete a resistance training workout comprised of barbell back squat, barbell bench press, and barbell conventional deadlift following either consuming breakfast and lunch, or the same amount of food consumed solely at lunch. For each testing session the participants will be provided with all food to consume prior to arriving at the laboratory. Major performance outcomes will be total repetition volume completed for each exercise (i.e. bench press, squat, and deadlift) and the entire workout (each individual trial), along with barbell kinematics for each exercise.

Participants will report to the laboratory on three separate occasions, with 3 to 10 days between each visit. At the first visit, after initial screening and provision of informed consent, each participant will undergo a performance screening and familiarization session to confirm eligibility and become accustomed to the study procedures. This familiarization session will include initial assessments of bench press, barbell back squat, and conventional deadlift maximal strength in order to determine final eligibility. Additionally, body composition will be assessed via dual-energy X-ray absorptiometry and digital anthropometry at this session for descriptive purposes. Following the familiarization session, each participant will complete two laboratory visits consisting of completion of the resistance training workout described below after consuming the provided meals either divided between breakfast and lunch (~3-4 hours after breakfast), or solely at lunch. This will ensure each participant consumes identical quantities and types of foods prior to both exercise sessions. Thus, the only difference will be the food distribution as two meals (breakfast and lunch) or one meal (lunch). Throughout the study, participants will be asked to maintain their normal lifestyle practices. In addition, participants will report their dietary intake during the 24-hour period prior to the first testing session and will be asked to replicate this intake during the 24-hour period prior to the subsequent testing sessions. A background questionnaire will also be completed to assess general supplement use.

PURPOSE

The purpose of this investigation is to examine the effect of breakfast consumption or omission on afternoon resistance training performance in habitual breakfast consumers and non-consumers.

GENERAL HYPOTHESIS

It is hypothesized that afternoon resistance training performance will be impaired in habitual breakfast consumers when breakfast is omitted, but similar decrements will not be observed in habitual non-consumers.

HYPOTHESES TO BE TESTED/SPECIFIC AIMS

Specific Aim 1. To determine the effect of breakfast consumption on afternoon resistance training performance.

Hypothesis. It is hypothesized that afternoon resistance training performance will not be impacted by breakfast consumption or omission when the cohort is examined as a whole.

Specific Aim 2. To determine whether habitual breakfast consumption patterns impact afternoon resistance training performance following consumption or omission of breakfast.

Hypothesis. It is hypothesized that habitual breakfast consumption patterns will impact the effect of breakfast consumption on resistance training performance. More specifically, performance will be negatively affected by the omission of breakfast in those who habitually consume breakfast. Yet the omission of breakfast will not negatively impact resistance training performance in those that regularly do not consume breakfast.

Specific Aim 3. To determine the impact of breakfast consumption on subjective responses throughout an afternoon resistance training session.

Hypothesis. It is hypothesized that subjective responses during afternoon resistance training will not be impacted by breakfast consumption or omission when the cohort is examined as a whole.

Specific Aim 4. To determine whether habitual breakfast consumption patterns influence subjective responses throughout an afternoon resistance training session, following consumption or omission of breakfast.

Hypothesis. It is hypothesized that worsened subjective responses will be observed after breakfast omission only in those who habitually consume breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* Body mass between 50 - 110 kg (110-242 lb)
* Generally healthy (defined as an absence of any disease or medical condition which could potentially be negatively affected by consumption of the commercially available dietary supplements or performance of exercise, including but not limited to musculoskeletal or cardiovascular diseases).
* Resistance-trained, defined as completing 2+ resistance training sessions per week for at least three months prior to screening.
* Participants must self-report either consuming or skipping breakfast ≥ 5 times per week for three months prior to screening.
* Participants must have reported regular training of the lower body through a multi-joint exercise such as the squat or leg press at least once weekly during the three-month period prior to screening.
* Participants must have reported regular training of the bench press or chest press variation at least once weekly during the three-month period prior to screening.
* Participants must have reported regular training of the deadlift or deadlift variation at least once weekly during the three-month period prior to screening.
* Female participants will be required to bench press ≥ 0.5 x body mass, barbell back squat ≥ 0.75 x body mass, and deadlift ≥ 1.0 x body mass to be eligible or this study.
* Male participants will be required to bench press ≥ 1.0 x body mass, barbell back squat ≥ 1.375 x body mass, and deadlift ≥ 1.75 x body mass to be eligible or this study.

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria.
* Pregnant or breastfeeding (for female participants)
* Taking prescription medication which could reasonably make participation unsafe for the participant or influence study outcomes
* An inability to complete resistance exercise due to injury or medical condition
* Inability to complete a 16 hour fast.
* Allergy to any of the ingredients in the provided breakfast and lunch.
* Current use of anabolic steroids
* Presence of a pacemaker or other implanted electrical device.
* Inability to perform the exercises with safe and proper form as determined by members of the research team.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Total Repetition Volume | 1 hour
  The total number of repetitions completed across four sets of the barbell back squat exercise, four sets of the barbell bench press exercise, and four sets of the conventional barbell deadlift exercise.
Squat Repetition Volume | 20 minutes
  The total number of repetitions completed across four sets of the barbell back squat exercise.
Bench Press Repetition Volume | 20 minutes
  The total number of repetitions completed across four sets of the barbell bench press exercise.
Deadlift Repetition Volume | 20 minutes
  The total number of repetitions completed across four sets of the conventional barbell deadlift exercise.
Average Concentric Barbell Velocity for Squat | 20 minutes
  The average barbell velocity during the concentric portion of the squat exercise across all repetitions.
Average Concentric Barbell Velocity for Bench Press | 20 minutes
  The average barbell velocity during the concentric portion of the bench press exercise across all repetitions.
Average Concentric Barbell Velocity for Deadlift | 20 minutes
  The average barbell velocity during the concentric portion of the deadlift exercise across all repetitions.
Peak Concentric Barbell Velocity for Squat | 20 minutes
  The peak barbell velocity during the concentric portion of the squat exercise across all repetitions.
Peak Concentric Barbell Velocity for Bench Press | 20 minutes
  The peak barbell velocity during the concentric portion of the bench press exercise across all repetitions.
Peak Concentric Barbell Velocity for Deadlift | 20 minutes
  The peak barbell velocity during the concentric portion of the deadlift exercise across all repetitions.
Average Power for Squat | 20 minutes
  The average power during the squat exercise across all repetitions.
Average Power for Bench Press | 20 minutes
  The average power during the bench press exercise across all repetitions.
Average Power for Deadlift | 20 minutes
  The average power during the deadlift exercise across all repetitions.
Peak Power for Squat | 20 minutes
  The peak power during the squat exercise across all repetitions.
Peak Power for Bench Press | 20 minutes
  The peak power during the bench press exercise across all repetitions.
Peak Power for Deadlift | 20 minutes
  The peak power during the deadlift exercise across all repetitions.

SECONDARY OUTCOMES:
Hunger | 1 hour
  Subjective rating of hunger as assessed by visual analog scale.
Desire to Eat | 1 hour
  Subjective rating of desire to eat as assessed by visual analog scale.
Fullness | 1 hour
  Subjective rating of fullness as assessed by visual analog scale.
Energy | 1 hour
  Subjective rating of energy as assessed by visual analog scale.
Focus | 1 hour
  Subjective rating of focus as assessed by visual analog scale.
Fatigue | 1 hour
  Subjective rating of fatigue as assessed by visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided